CLINICAL TRIAL: NCT06972927
Title: VertiGreens Investigating the Effects of Iron Biofortification of Microgreens on Iron Status in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 821
Record Dates: First submitted 2025-05-06; First posted 2025-05-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Iron Biomarkers/Status
Keywords: vertical farming; iron biomarkers; iron status; biofortification; microgreens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vertigreens (Experimental): Phase 1: Habitual diet (1 week) Phase 2: Vertigreens diet: One smoothie a day containing biofortified microgreens (4 weeks)
  Interventions: Other: Smoothie containing iron biofortified microgreens

INTERVENTIONS:
Other: Smoothie containing iron biofortified microgreens — 30g of iron biofortified microgreens consumed within a smoothie for 28 days

SUMMARY:
The investigators present a diet intervention study, to be conducted as a within-subject design, to assess the effect of the provision of iron biofortified microgreens on iron intake and status in women of reproductive age and postmenopausal women. This will be investigated by providing smoothie kits for 28 days containing these microgreens and determining the impact on iron biomarkers. The investigators will also assess habitual diet, BMI, physical activity and gastrointestinal symptoms. This study will be a proof-of-concept exploratory study to explore diet based biofortification through vertical farming systems.

DETAILED DESCRIPTION:
In this study microgreens that were grown using agronomic iron biofortification will be supplied to women to add to their diet to establish the potential nutritional impact of iron biofortified microgreens on overall iron intake and iron status. Furthermore, it will assess the adherence to the provided consumption recommendations of the biofortified crops.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females
* 15 of reproductive age (18-49)
* 15 postmenopausal (not had their period for an entire year)

Exclusion Criteria:

Medication exclusion criteria:

* Supplementing iron or vitamin B12
* Smoking or vaping
* Taking anticoagulant medication (blood thinners) except for Aspirin 75mg

Medical exclusion criteria:

* Anyone who is planning to be pregnant, is pregnant or breastfeeding
* Anyone with iron or vitamin B12 deficiency anaemia
* Anyone with history of anaemia in the past 3 months that required treatment
* Anyone who has Hb <120 g/L (12 g/dL) at screening
* Anyone with food allergies, self-reported food sensitivity or intolerance
* Anyone with coeliac disease or gluten intolerance
* Anyone suffering from a psychiatric disorder or any type of substance abuse
* Anyone with Type 1 diabetes and Type 2 diabetes
* Anyone suffering from unregulated thyroid disease
* Anyone with gastrointestinal conditions or bariatric surgery
* Anyone with haematological conditions including Thrombocytopaenia and Sickle cell anaemia

Other exclusion criteria:

* Anyone with unsuitable veins for blood sampling
* Anyone who donated blood in the last 16 weeks
* Anyone who is unable to fluently speak, read and understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Haemoglobin status change from baseline | Measured at study day 1 and on study day 28
  Iron status changes in haemoglobin
Serum iron status change from baseline | Measured at study day 1 and on study day 28
  Iron status changes in serum iron
Ferritin status change from baseline | Measured at study day 1 and on study day 28
  Iron status changes in ferritin
CRP change from baseline | Measured at study day 1 and on study day 28
  Changes in CRP
Dietary iron intake changes compared to habitual diet | every study day (28 days)
  Dietary iron intake changes in iron intake compared to habitual diet measured though food diaries

SECONDARY OUTCOMES:
Serum Vitamin B12 status change from baseline | Measured on study day 1 and on study day 28
  Vitamin B12 status changes
Adherence to consumption of microgreens/smoothie | every study day (28 days)
  intake measured through food diaries

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Johnstone, Prof, Principal Investigator — University of Aberdeen, Rowett Institute of Nutrition and Health
Locations (1):
- Rowett Institute, University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No